CLINICAL TRIAL: NCT06614543
Title: Feasibility Testing of Plant-Based Meal Replacement Products Made With Manitoba Crop Ingredients for Weight Loss and Diabetes Remission
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Seven Oaks Hospital Chronic Disease Innovation Centre (Network); The Wellness Institute (Unknown); Sustainable Canadian Agricultural Partnership (Unknown)
Responsible Party: Principal Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS26095 (B2023:073)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Weight Loss; Prediabetes; Diabetes
Keywords: Weight Loss Clinic; Meal Replacement
MeSH Terms: conditions — Weight Loss; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The WLC program plus meal replacements (Active Comparator): Participants will have a choice on what type of meal replacement they will consume each day (either a bar or a shake) and will record this in the product consumption log.
  Interventions: Dietary Supplement: Meal Replacement
- The WLC program only (No Intervention)

INTERVENTIONS:
Dietary Supplement: Meal Replacement — These meal replacements provide plant-based protein, fibre and fatty acids that have been shown to have health benefits related to chronic disease.
  Arms: The WLC program plus meal replacements

SUMMARY:
The goal of this clinical trial is to advance the development of the WI meal replacements by evaluating the acceptance and feasibility of the meal replacements within the Wellness Institute's Weight Loss Clinic program (WLC). The main questions it aims to answer are:

* To determine whether the incorporation of WI meal replacements into their weight loss clinic design is feasible.
* To determine whether weight loss is supported by a plant-based meal replacement.
* To assess efficacy of the meal replacements by measuring changes in lifestyle behaviours and risk factors for chronic disease compared to non-meal replacement weight loss program members.
* To assess remission of diabetes and pre-diabetes.

Researchers will compare the WLC program plus meal replacements to the WLC program without the meal replacements to evaluate the implementation of the meal replacements into the WLC.

Participants will follow their WLC program for 16 weeks, and those in the intervention group will begin their meal replacements. Participants will have a choice on what type of meal replacement they will consume each day (either a bar or a shake) and will record this in the product consumption log.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or above
* Live within the province of MB
* Ability to give written informed consent in English.
* Enrolled in the Wellness Institute Weight Loss Clinic

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the program.
* Participants with known allergies to the meal replacement ingredients
* Has an active eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of incorporating the WI meal replacements into their weight loss clinic design. | At Enrollment (Week 0) and End of Study (Week 16)
  Feasibility will be demonstrated if the following five criteria are met:
  1. Eligibility to randomization ratio is greater than 0.5, calculated as the ratio of individuals within the WI WLC program who were randomized to the trial to the number eligible to participate who were approached to participate.
  2. The percentage of participants who complete the 16-week program in the meal replacement arm is equivalent (plus or minus 10%) or greater than the standard arm.
  3. Follow up of greater than 85% of participant outcomes.
  4. Adherence to the meal replacement intervention calculated by consumption of greater than 75% dispensed products as documented in the Product Consumption Log
  5. Product Acceptability using an Exit Questionnaire consisting of a 9-point hedonic box scale to assess mean acceptability values of 6 or greater (like at least slightly) in 75% or more of the participants.

SECONDARY OUTCOMES:
Changes in Body Weight | At Enrollment (Week 0) and End of Study (Week 16)
  Body weight will be measured in kg to the nearest 0.1 kg by an exercise professional.
Changes in Waist Circumference | At Enrollment (Week 0) and End of Study (Week 16)
  Waist circumference in cm will be measured to the nearest 0.1 cm at the umbilicus, between the last rib and iliac crest using a fibreglass tape measured by an exercise professional.
Changes in BMI | At Enrollment (Week 0) and End of Study (Week 16)
  Body Mass Index will be calculated using the formula BMI = kg/m2; where kg is the weight in kilograms and m2 is height in metres squared.
Cardiovascular Assessment | At Enrollment (Week 0) and End of Study (Week 16)
  Using the Framingham Risk Score, cardiovascular risk will be calculated based on age, HDL-C, total cholesterol, systolic blood pressure, smoking status, and diabetes status to determine the participant's 10-year risk of cardiovascular disease and identification of metabolic syndrome.
Changes is Quality of Life | At Enrollment (Week 0) and End of Study (Week 16)
  Quality of life will be measured through the SF-36 quality of life questionnaire. The SF-36 measures nine areas: physical functioning, role functioning (emotional), role functioning (physical), energy/fatigue, emotional well-being, social functioning, pain, general health, and health change. A higher score indicates greater levels of quality of life.
Changes in Medication | At Enrollment (Week 0) and End of Study (Week 16)
  Changes in medications, dose, unit and frequency will be captured to assess remission of diabetes and pre-diabetes.
Changes in HemaglobinA1C | At Enrollment (Week 0) and End of Study (Week 16)
  Changes in hemaglobinA1C will be used to assess remission of diabetes and pre-diabetes. Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the hemoglobin A1C as a percentage according to their established protocols.

OTHER OUTCOMES:
Changes in Systolic Blood Pressure | At Enrollment (Week 0) and End of Study (Week 16)
  Systolic blood pressure in mmHg is measured in triplicate, on the non-dominant arm in a sitting position by an exercise professional using a validated oscillometric blood pressure monitor.
Changes in Diastolic Blood Pressure | At Enrollment (Week 0) and End of Study (Week 16)
  Diastolic blood pressure in mmHg is measured in triplicate, on the non-dominant arm in a sitting position by an exercise professional using a validated oscillometric blood pressure monitor.
Changes in Heart Rate | At Enrollment (Week 0) and End of Study (Week 16)
  Heart rate in beats per minute is measured in triplicate, on the non-dominant arm in a sitting position by an exercise professional using a validated oscillometric blood pressure monitor.
Changes in Physical Activity | At Enrollment (Week 0) and End of Study (Week 16)
  Measured using the International Physical Activity Questionnaire - Short Form - (IPAQ-S)
Change in Physical Activity Behaviour Patterns | At Enrollment (Week 0) and End of Study (Week 16)
  Assessed using total active minutes per day as measured by multi-directional accelerometry for 5 days. Participants will be asked to wear the accelerometer at all times.
Changes in Dietary Intake Behaviours | At Enrollment (Week 0) and End of Study (Week 16)
  Dietary intake behaviours will be measured through The Mindful Eating Questionnaire. The Mindful Eating Questionnaire recognizing patterns of overeating or eating in response to stress, boredom, or other emotions. Scoring is based on five categories, which include Awareness (being aware of how food looks, tastes and smells); Distraction (focusing on other things while eating); Disinhibition (eating even when full); Emotional Response (eating in response to sadness or stress); and External Cues (eating in response to environmental cues, such as advertising)
Changes in Dietary Intake Behaviours | At Enrollment (Week 0) and End of Study (Week 16)
  Changes in dietary intake behaviours will be measured through the Three Factor Eating Questionnaire which is comprised of 18 items, measuring uncontrolled eating, restrained eating and emotional eating. The higher the score represents more dependency to cognition, stress or emotion the eating patterns.
Changes in Dietary Intake - Number of Meals | At Enrollment (Week 0) and End of Study (Week 16)
  Number of meals will be captured with a meal being defined as food intake greater than 500 kcal. Dietary intake will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Dietary Intake - Number of Snacks | At Enrollment (Week 0) and End of Study (Week 16)
  Number of snacks will be captured with a meal being defined as food intake less than 500 kcal. Dietary intake will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Dietary Intake - Energy | At Enrollment (Week 0) and End of Study (Week 16)
  Energy will be measured in kCals and will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Dietary Intake - Protein | At Enrollment (Week 0) and End of Study (Week 16)
  Protein will be measured in grams and will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Dietary Intake - Fat | At Enrollment (Week 0) and End of Study (Week 16)
  Fat will be measured in grams and will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Dietary Intake - Available Carbohydrates | At Enrollment (Week 0) and End of Study (Week 16)
  Available carbohydrates will be measured in grams and will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Dietary Intake - Fibre | At Enrollment (Week 0) and End of Study (Week 16)
  Fibre will be measured in grams and will be captured using the RxFood app. RxFood is a type of AI-driven, image based dietary assessment tool that has already demonstrated clinical benefits in various adult and pediatric clinical settings and in research as a data collection tool. Strong correlation and strength of agreement have been illustrated between RxFood and nutrient estimates from Esha's Research Nutrition analysis software, which is an industry choice for nutritional analysis and regulatory compliance (Jefferson et al, 2020).
Changes in Sleep Patterns | At Enrollment (Week 0) and End of Study (Week 16)
  An ActiGraph activity monitor will be used to measure sleep quality patterns for 5 days, with participants asked to wear the monitor at all times, including when they sleep.
Changes in Total Cholesterol | At Enrollment (Week 0) and End of Study (Week 16)
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.
Changes in High density lipoprotein cholesterol | At Enrollment (Week 0) and End of Study (Week 16)
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.
Changes in Low density lipoprotein cholesterol | At Enrollment (Week 0) and End of Study (Week 16)
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.
Changes in Triglycerides | At Enrollment (Week 0) and End of Study (Week 16)
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.
Changes in Total Cholesterol and High-Density Lipoprotein Cholesterol Ratio | At Enrollment (Week 0) and End of Study (Week 16)
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.
Changes in Hemoglobin A1C | At Enrollment (Week 0) and End of Study (Week 16)
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Dylan MacKay, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Seven Oaks Hospital Chronic Disease Innovation Centre, Winnipeg, Manitoba, Canada